CLINICAL TRIAL: NCT05915442
Title: Phase II Single Arm Study Testing SBRT, Adenosine Signaling Modulation (AB680, AB928), and Immune Checkpoint Inhibition (AB122) for Men With Hormone Sensitive Oligometastatic Prostate Cancer
Brief Title: Adenosine Signaling Modulation and Immune Checkpoint Inhibition With Hormone Sensitive Oligometastatic Prostate Cancer
Acronym: SBRT-AMICO
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Catherine Spina (Other)
Collaborators: Arcus Biosciences, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Catherine Spina, Assistant Professor of Radiation Oncology, Columbia University
Organization: Columbia University (Other)
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: AAAU4675
Record Dates: First submitted 2023-06-07; First posted 2023-06-23 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Oligometastatic Prostate Cancer
Keywords: Adenosine Signaling; AB680; AB928; AB122; Quemliclustatm; Etrumadenant; Zimberelimab
MeSH Terms: interventions — quemliclustat; zimberelimab; Radiosurgery

STUDY DESIGN:
Intervention Model Description: Simon Two-Stage design: In the first stage, trial will enroll 14 patients. If two or more patients show progression at 6 months, the study is terminated at the end of stage I. However, if 13 of the 14 remain free from progressive disease at 6 months, then the study would move onto the second stage. In this stage, n=9 additional patients will be enrolled, for a total of 23 total. If 21 of the 23 patients remain progression-free at 6 months, then the null hypothesis is rejected, and we will consider the addition of quemliclustat, etrumadenant, and zimberelimab to SBRT worthy of further study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment with quemliclustatm, etrumadenant, zimberelimab and SBRT (Experimental): Subjects with metastatic prostate cancer will receive quemliclustat and etrumadenant for 4 weeks prior to metastasis-directed SBRT (Stereotactic Body Radiation Therapy). Within one week of completing SBRT, subjects will also start zimberelimab.
  Interventions: Drug: Quemliclustat; Drug: Etrumadenant; Drug: Zimberelimab; Radiation: Stereotactic Body Radiation Therapy

INTERVENTIONS:
Drug: Quemliclustat — 100mg IV once every two weeks
  Other Names: AB680
Drug: Etrumadenant — 150 mg orally (PO) once a day (QD)
  Other Names: AB928
Drug: Zimberelimab — 240 mg IV once every two weeks starting within 1 week of completing metastasis-directed SBRT
  Other Names: AB122
Radiation: Stereotactic Body Radiation Therapy — Standard of care metastasis-directed hypofractionated radiotherapy treatment starting 4 weeks (+/- 1 week) of starting Etrumadenant and Quemliclustat
  Other Names: SBRT

SUMMARY:
This study will evaluate the safety and effectiveness of a combination of study drugs including zimberelimab, etrumadenant, and quemliclustat in combination with metastasis-directed irradiation in men with hormone sensitive oligometastatic prostate cancer.

The study aims to test the hypothesis that targeted inhibition of the adenosine signaling axis (quemliclustat (CD73 antagonist) + etrumadenant (A2AR/A2BR antagonist)) and immune checkpoint inhibition (zimberelimab, α-PD-1) in combination with metastasis-directed stereotactic body radiation therapy (SBRT) will improve local control, progression-free survival (PFS), and hormone therapy-free survival and mitigate immunosuppressive changes to the tumor microenvironment (TME), compared to SBRT alone.

DETAILED DESCRIPTION:
The optimal therapeutic approach to men with oligometastatic (1-3 or 1-5 sites of metastatic disease) prostate cancer is ever more important as advanced imaging technologies are becoming standard of care, providing clinicians with the tools to accurately diagnose and localize oligometastatic prostate cancer. Hence, methods to improve the local curative potential of stereotactic body radiation therapy (SBRT) is a timely and important opportunity. In addition, previous data suggest that the adenosine A2A pathway may be a particularly attractive avenue for intervention in the context of radiation, thus influencing multiple suppressive populations within the tumor microenvironment (TME).

Immunotherapy based on the PD-1/PD-L1 signaling axis is a mainstay of therapy across multiple types of malignancies. This study aims to evaluate the effectiveness of a PD-1 inhibitor (zimberelimab) in combination with a selective dual antagonist of A2aR and A2bR (etrumadenant) and an anti-CD73 (quemliclustat). Immune checkpoint inhibitors and targeted inhibitors of the adenosine signaling axis modulate the TME and aspects of the systemic immune system to overcome tumor-induced immune suppression and improve responses to therapy.

This study aims to determine the effect of etrumadenant, quemliclustat and zimberelimab [experimental] when given with ablative radiation (SBRT)[standard of care] on the oligoprogressive disease (hormone sensitive oligometastatic prostate cancer), defined by being free from radiographic progression of irradiated target metastases and PSA (prostate surface antigen) response at 6 months. PSA response, local control, progression-free survival (PFS), treatment response, ADT-free survival, time-to-pain, and safety and tolerability will also be measured. By employing a Simon Two-Stage design, the trial will test whether or not etrumadenant + quemliclustat and zimberelimab combined with ablative radiation (SBRT) will improve PFS compared to SBRT alone (ORIOLE).

ELIGIBILITY:
Inclusion Criteria:

1. Patient must have histologically confirmed adenocarcinoma of the prostate.
2. Patient's primary prostate cancer tumor treated with surgery and/or radiation (+/- ADT).
3. Patients must have one to three asymptomatic metastatic tumors of the bone or soft tissue that developed in the preceding 6 months that are < 5cm or < 250 cm3.
4. Prostate-specific antigen (PSA) > 0.5 ng/mL but < 50ng/ml
5. PSA doubling time (PSADT) < 15 months (using all available PSA values from time of relapse)
6. Testosterone > 125 ng/mL
7. Age ≥18 years.
8. Patient must have life expectancy > 12 months.
9. Eastern Cooperative Oncology Group (ECOG) performance status 0-2
10. Normal organ and marrow function as defined below:

    * leukocytes ≥3,000/mcL
    * absolute neutrophil count ≥1,500/mcL
    * platelets ≥100,000/mcL
    * total bilirubin within normal institutional limits
    * aspartate transaminase (AST)(serum glutamic-oxaloacetic transaminase (SGOT))/alanine transaminase (ALT)(serum glutamic-pyruvic transaminase (SGPT) ) ≤2.5 × institutional upper limit of normal creatinine, within normal institutional limits
11. Male participants with female partners of childbearing potential are required to use highly effective contraceptive measures which include condom use. A man is considered fertile after puberty unless permanently sterile by bilateral orchidectomy. A female partner of is considered a woman of childbearing potential (WOCBP) following menarche and until becoming postmenopausal unless permanently sterile.

    * Permanent sterilization methods include hysterectomy, bilateral salpingectomy and bilateral oophorectomy.
    * A postmenopausal state is defined as no menses for 12 months without an alternative medical cause. A high follicle-stimulating hormone (FSH) level in the postmenopausal range may be used to confirm a postmenopausal state in women not using hormonal contraception or hormonal replacement therapy. However, in the absence of 12 months of amenorrhea, a single FSH measurement is insufficient.

    Highly effective contraceptive measures include:
    * Combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation: oral, intravaginal, transdermal
    * Progestogen only hormonal contraception associated with inhibition of ovulation: oral, injectable, implantable
    * Intrauterine device
    * Intrauterine hormone-releasing system
    * Surgical sterilization
    * The male participant is vasectomized (with documented medical confirmation of surgical success) and is the sole sexual partner of the WOCBP participant
    * Female partner of the male participant has undergone bilateral tubal ligation
    * Complete sexual abstinence defined as refraining from heterosexual intercourse during the entire period of risk associated with study treatment. The reliability of sexual abstinence needs to be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the participant.
12. Male participants should refrain from donating sperm for 180 days after the last dose of the study drugs.
13. Patient must have the ability to understand and the willingness to sign written informed consent.

Exclusion Criteria:

1. Patient may not have had prior systemic therapy, with the exception of androgen deprivation therapy (ADT) associated with treatment of the primary prostate tumor or with salvage radiation therapy. The ADT could not exceed 3-years in duration and must have occurred greater than 6 months before time of enrollment.
2. Patients with known brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events.
3. Spinal cord compression or impending spinal cord compression.
4. Pulmonary and/or liver metastases > 1.0cm in largest dimension.
5. History of malignancy other than prostate cancer within 2 years prior to screening, except for malignancies with a negligible risk of metastasis or death (e.g., 5-year OS rate > 90%), such as nonmelanoma skin carcinoma or ductal carcinoma in situ.
6. Use of other investigational agents or treatment protocol.
7. Treatment with therapeutic oral or intravenous (IV) antibiotics within 2 weeks prior to initiation of study treatment with the exception of patients receiving prophylactic antibiotics (e.g., to prevent a urinary tract infection or chronic obstructive pulmonary disease exacerbation) are eligible for the study.
8. Inability to swallow medications.
9. Malabsorption condition that would alter the absorption of orally administered medications.
10. Grade ≥ 3 hemorrhage or bleeding event within 28 days prior to initiation of study treatment.
11. History of idiopathic pulmonary fibrosis, organizing pneumonia (e.g., bronchiolitis obliterans), drug induced pneumonitis, or idiopathic pneumonitis, or evidence of active pneumonitis on screening chest computed tomography (CT) scan.
12. Severe infection within 4 weeks prior to initiation of study treatment, including, but not limited to, hospitalization for complications of infection, bacteremia, or severe pneumonia.
13. Positive total hepatitis B core antibody (HBcAb) test at screening. Patients can be eligible if positive total HBcAb test followed by a negative hepatitis B virus (HBV) DNA test at screening. The HBV test will be performed only for participants who have a positive total HBcAb test. Due to safety concerns related to viral activation, development of a secondary malignancy, as well as the potential for increased treatment-related toxicity, eligible participants must not have evidence of chronic viral infection at screening.
14. Due to the potential risk for drug-drug interactions with etrumadenant, participants must not have had:

    1. Oral treatment with strong inhibitors of breast cancer resistance protein (BCRP) (e.g., cyclosporin A, eltrombopag) or BRCP substrates with a narrow therapeutic window, administered orally (e.g., prazosin, rosuvastatin) within 4 weeks or 5 drug-elimination half-lives of the drug (whichever is longer) prior to initiation of study treatment.
    2. Oral treatment with strong inhibitors of P-glycoprotein (P-gp) substrates (e.g., itraconazole, quinidine, verapamil, dronedarone, ranolazine) or P-gp with a narrow therapeutic window, administered orally (e.g., digoxin) within 4 weeks or 5 drug-elimination half-lives of the drug (whichever is longer) prior to initiation of study treatment.
    3. Treatment with known strong CYP3A4 inducers (e.g., rifampin, phenytoin, carbamazepine, phenobarbital, and St. John's Wort) or strong CYP3A4 inhibitors (e.g., clarithromycin, grapefruit juice, itraconazole, ketoconazole, posaconazole, telithromycin, and voriconazole) within 4 weeks or 5 half-lives of the drug (whichever is longer) prior to initiation of study treatment.
    4. Treatment with known strong UDP-glucuronosyltransferases (UGTs) of UGT1A1, 1A4, 1A9 and 2B4 inhibitors (e.g., atazanavir) within 4 weeks or 5 half-lives of the drug, whichever is longer, prior to the initiation of study treatment.
    5. Treatment with known sensitive substrates of BSEP within 4 weeks or 5 half-lives of the drug, whichever is longer, prior to the initiation of study treatment.
    6. Treatment with known sensitive substrates of OCT2 within 4 weeks or 5 half-lives of the drug, whichever is longer, prior to the initiation of study treatment.
    7. Treatment with known sensitive substrates of MATE1 within 4 weeks or 5 half-lives of the drug, whichever is longer, prior to the initiation of study treatment.
15. Immunosuppression (e.g., solid organ transplant on immunosuppression).
16. No known HIV, or active with Hepatitis C Virus (HCV) or Hepatitis B Virus (HBV).
17. Active autoimmune disease.
18. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
19. Inability to lie flat to tolerate computed tomography (CT) simulation study and oligometastasis-directed stereotactic body radiotherapy (SBRT).
20. Use of any live vaccines against infectious diseases within 28 days of first dose of investigational products.
21. Refusal to sign informed consent.

Ages: 18 Years to 99 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Biochemical recurrence-free survival at 12-months | 12 months
  Biochemical recurrence is defined as a 0.2 ng/ml increase in PSA above the post-SBRT PSA nadir. Patient will be followed until biochemical recurrence, death, or end of study, whichever comes first. Patients who are alive and biochemical recurrence free will be censored at the last PSA measurement date.

SECONDARY OUTCOMES:
Biochemical recurrence-free survival at 6-months | 6 months
  To estimate the proportion of men treated with quemliclustat + etrumadenant + zimberelimab + SBRT who are free from biochemical failure at 6-months.
To estimate treatment response based on CT at 6-months | 6 months
  Report the percentage of patients with PD, CR, PR, and SD based on CT imaging among patients treated with oligometastasis-directed SBRT + quemliclustat + etrumadenant + zimberelimab at 6-months.
To estimate treatment response based on nuclear bone scan at 6-months. | 6-months
  Report the percentage of patients with PD, CR, PR, and SD based on nuclear bone scan among patients treated with oligometastasis-directed SBRT + quemliclustat + etrumadenant + zimberelimab at 6-months.
To estimate treatment response based on PSMA-PET scan at 6-months. | 6-months
  Report the percentage of patients with PD, CR, PR, and SD based on PSMA-PET scan among patients treated with oligometastasis-directed SBRT + quemliclustat + etrumadenant + zimberelimab at 6-months.
Proportion of patients who start ADT. | 6, 12 months and 3 years.
To estimate pain over time. | Every 12 weeks for 3.5 years
  Quantify pain using a numeric 10-point scale using the Brief Pain Inventory (BPI) every 12 weeks from time of enrollment.
To assess the safety and tolerability of oligometastasis-directed SBRT + quemliclustat + etrumadenant + zimberelimab. | 6, 12 months and 3 years
  Adverse events graded by CTCAE v5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Catherine S. Spina, MD, PhD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Irving Medical Center / NewYork-Presbyterian Hospital, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No